CLINICAL TRIAL: NCT00625820
Title: Safety and Efficacy of Tetrahydrobiopterin in Patients With Chronic Kidney Disease (CKD) and Albuminuria: An Open-Label Pilot Study
Brief Title: Tetrahydrobiopterin in Patients With Chronic Kidney Disease (CKD) and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Rajiv Saran, MD, MS, MRCP, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00016705
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Disease; Albuminuria
Keywords: Kidney Disease; Albuminuria; Glomerular filtration rate
MeSH Terms: conditions — Kidney Diseases; Albuminuria | interventions — phenoptin; sapropterin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6R BH4 (Experimental): Subjects will receive 6R-BH4 400mg bid for 6 weeks, sequentially followed by 6R-BH4 plus Vitamin C 500mg bid for another 6 weeks. Patients will have scheduled visits at Weeks 0,3,6,9 and 12, with an exit-visit at week 16. Albuminuria will be assessed in 24-hour urine collections as well as early morning spot urine samples for albumin:creatinine ratio. Blood and urine will be tested for routine clinical laboratory tests, blood nitric oxide (NO), and also archived for later assays for special biomarkers. The primary outcome will be level of albuminuria as measured in a 24-hour urine collection at 6 and 12 weeks of therapy. Secondary outcomes will include urine albumin/creatinine ratio, estimated glomerular filtration rate (eGFR), and blood pressure .
  Interventions: Drug: 6R BH4; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: 6R BH4 — 400 mg 6R BH4 oral BID for 6 weeks then 400 mg of 6R BH4 for another 6 weeks in all arms
  Other Names: Tetrahydrobiopterin
Dietary Supplement: Vitamin C — 500 mg Vitamin C oral BID for another 6 weeks

SUMMARY:
Patients with chronic kidney disease (CKD) and albuminuria are at increased risk of developing cardiovascular disease (CVD) which is often associated with hypertension, left ventricular hypertrophy, endothelial dysfunction and increased generation of reactive oxygen species (ROS). These patients also manifest a decrease in nitric oxide (NO) availability which is thought to play an important role in their progressive vascular disease.

Tetrahydrobiopterin (BH4), an essential cofactor for endothelial nitric oxide synthase(eNOS), an important regulator of NO and that is a key mediator of endothelial dysfunction. Changes in NO availability are believed to contribute to endothelial dysfunction seen in CKD and common CVD states. 6R-tetrahydrobiopterin (6R-BH4 or sapropterin dihydrochloride) is an investigational oral drug that is being evaluated to determine whether it will restore NO availability, leading to beneficial effects on vascular function and ultimately positive clinical outcomes in patients with CKD. The primary endpoint in this study is the level of albuminuria, an easily measured marker that has served as a predictor of kidney disease progression. If 6R-BH4 reduces albuminuria in patients with kidney disease, it may have implications to slow the disease progression as well as decreased risk of CVD.

DETAILED DESCRIPTION:
ABSTRACT Background: Chronic kidney disease (CKD) is characterized by a high propensity to cardiovascular disease (CVD); therefore treatments that impact both CKD and CVD are needed. CKD is accompanied by endothelial dysfunction and nitric oxide (NO) deficiency. Tetrahydrobiopterin (BH4), an important co-factor for endothelial NO synthase (eNOS) increases the availability of NO. Administration of BH4 has the potential to improve endothelial function and thereby reduce albuminuria in CKD.

Patients and Methods: This Phase 2 open-label study is designed to assess the efficacy and safety of twice daily oral dosing of 6R-BH4 in 30 subjects with CKD (estimated glomerular filtration rate (eGFR) ≥40ml/min/1.73m2).

Trial Design: Subjects will receive 6R-BH4 400mg bid for 6 weeks, sequentially followed by 6R-BH4 plus Vitamin C 500mg bid for another 6 weeks. Patients will have scheduled visits at Weeks 0,3,6,9 and 12, with an exit-visit at week 16. Albuminuria will be assessed in 24-hour urine collections as well as early morning spot urine samples for albumin:creatinine ratio. Blood and urine will be tested for routine clinical laboratory tests, blood NO, and also archived for later assays for special biomarkers. The primary outcome will be level of albuminuria as measured in a 24-hour urine collection at 6 and 12 weeks of therapy. Secondary outcomes will include urine albumin/creatinine ratio, eGFR, and blood pressure. Adverse events will be monitored closely.

Data analysis: For all patients combined and for each of the above outcomes, we will sequentially compare each time point to the baseline level using paired t-tests. For the comparison of 6R-BH4 versus 6R-BH4+vitamin C, we will compare albuminuria at 6 and 12-weeks, adjusted for baseline values, using regression analysis. We will also use regression to test for an interaction between baseline value and treatment group.

Anticipated results: We postulate that 6R-BH4 alone or in conjunction with high dose vitamin C will reduce albuminuria in patients with CKD by improvement in endothelial function that is integral to glomerular filtration.

Future Implications: Reduction in albuminuria if demonstrable, will have implications for simultaneous renal and cardiovascular protection. This will need to be confirmed in a larger randomized controlled clinical trial in subjects with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with controlled hypertension (blood pressure (BP) less than 150/90 mmHg) using standard antihypertensive medications.
* Stable chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) 40-90 ml/min/173m2 by the abbreviated Modification of Diet in Renal Disease (MDRD) equation and with a rate of decline of eGFR no greater than 1ml/min/1.73m2 per month over the prior 3 months with albuminuria (urine albumin excretion in the 24-hr urine sample of between 300-3000mg).
* No concomitant use with:

  * Vitamin C supplements
  * Multivitamins containing vitamin C
  * Any other dietary supplements, nutraceuticals, or other over-the- counter products containing vitamin C
  * Vitamin E containing supplements
* Concurrently taking study approved antihypertensive medications at a stable dose for at least 3 months prior to screening.
* Sexually active subjects must be willing and able to use an acceptable method of contraception
* Females of childbearing potential must have a negative pregnancy test at screening. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to screening, or who have had total hysterectomy.

Exclusion Criteria:

* Uncontrolled hypertension with BP greater than 150/90 or with frequent changes to antihypertensive regimen during the last 3 months.
* Concurrent disease or condition that would interfere with study participation or safety, such as bleeding disorders, history of syncope or vertigo; severe gastroesophageal reflux disease (GERD) or gastric ulcers; heart failure; symptomatic coronary or peripheral vascular disease; arrhythmia; serious neurologic disorders, including seizures; or organ transplant.
* Diabetics that are uncontrolled, unstable, newly diagnosed, or have undergone major changes in therapy in the last three months or HbA1C consistently greater than 9.0.
* Any severe comorbid condition that would limit life expectancy to less than 6 months.
* Advanced stage III CKD or worse , i.e. eGFR less than 40 ml/min/1.73m2 (by abbreviated MDRD formula).
* History of nephrolithiasis.
* Patients with albuminuria due to causes other than hypertension and /or diabetes; e.g., systemic lupus erythematosus (SLE).
* Hepatic enzyme concentrations greater than 2 times the upper limit of normal.
* HIV infection, hepatic cirrhosis, other preexisting liver disease, or positive HIV, Hepatitis B or C test at screening.
* Concomitant treatment with drugs known to inhibit folate metabolism, Levodopa, phosphodiesterase (PDE) 5 inhibitors or PDE 3 inhibitors.
* Myocardial infarction, stroke, or surgery within the last 60 days prior to screening.
* History of alcohol and/or drug abuse.
* Pregnant or breastfeeding at screening, or planning to become pregnant (subject or partner) at any time during the study.
* Previous treatment with tetrahydrobiopterin (6R-BH4).
* Has known hypersensitivity to 6R-BH4 or its excipients.
* Any condition that, in the view of the principal investigator (PI), places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saran, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from nephrology clinics based on baseline estimated glomerular filtration rate (eGFR). Informed consent was obtained from each patient prior to the study based on institutional review board (IRB) approved guidelines.
Pre-assignment Details: Seventeen patients were recruited and all started the trial.
Groups:
- 1BH4, BH4 + Vitamin C: N/A
  Tetrahydrobiopterin (6R BH4) : 400 mg 6R BH4 oral BID for 6 weeks then 400 mg of 6R BH4 for another 6 weeks
  Vitamin C : 500 mg Vitamin C oral BID for another 6 weeks
Period: Overall Study
Arm/Group | 1BH4, BH4 + Vitamin C
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 1BH4, BH4 + Vitamin C: NA
  Tetrahydrobiopterin (6R BH4) : 400 mg 6R BH4 oral BID for 6 weeks then 400 mg of 6R BH4 for another 6 weeks
  Vitamin C : 500 mg Vitamin C oral BID for another 6 weeks
Arm/Group | 1BH4, BH4 + Vitamin C
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is Level of Albuminuria.
Description: Early morning urine specimens were collected to calculate albumin and creatinine ratio (albuminuria) at 6 and 12 weeks of therapy.
Time Frame: 12 weeks
Population: All participants who finished the trial were analyzed
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1BH4, BH4 + Vitamin C
Number analyzed (Participants) | 16
ratio
  Albuminuria at week 6 | 927.9 (244.9)
  Albuminuria at week 12 | 897.1 (217.9)

2. Secondary Outcome: Systolic Blood Pressure Measured at 6 and 12 Weeks of Therapy.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | 1BH4, BH4 + Vitamin C
Number analyzed (Participants) | 16
mmHG
  Systolic Blood Pressure at week 6 | 143.1 (5.1)
  Systolic Blood Pressure at week 12 | 134.1 (3.71)

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Measured at 6 and 12 Weeks of Therapy.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | 1BH4, BH4 + Vitamin C
Number analyzed (Participants) | 16
ml/min/1.73m2
  eGFR at week 6 | 68.1 (6.7)
  eGFR at week 12 | 70.8 (6.4)

ADVERSE EVENTS:
Arm/Group | BH4, BH4 + Vit C
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BH4, BH4 + Vit C (N=17)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — One patient did develop kidney stones requiring stone extraction and lithotripsy after.

LIMITATIONS AND CAVEATS:
It was a small single center non-randomized pilot study & was not powered to detect significant changes in albuminuria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No